CLINICAL TRIAL: NCT00083174
Title: A Phase III Randomized Study of Exemestane Versus Placebo in Postmenopausal Women at Increased Risk of Developing Breast Cancer
Brief Title: Exemestane in Preventing Cancer in Postmenopausal Women at Increased Risk of Developing Breast Cancer
Acronym: ExCel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Grupo Espanol de Investigacion del Cancer de Mama (Other); UNICANCER (Other)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MAP3; CAN-NCIC-MAP3 (Registry Identifier: PDQ); PFIZER-EXEAPO-0028-150 (Other: Pfizer); CDR0000363802 (Other: PDQ); NCT00304486 (obsolete NCT alias)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Exemestane (Other): one 25 mg tablet daily in am
  Interventions: Drug: exemestane

INTERVENTIONS:
Drug: exemestane — one 25 mg tablet daily in am

SUMMARY:
RATIONALE: The MAP.3 study was designed to test whether hormone therapy using exemestane may prevent breast cancer by blocking the production of estrogen.

PURPOSE: The study protocol was amended in May 2011 and the current purpose of the study is to allow all study participants the opportunity to complete 5 years of exemestane.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

Previously: To determine if exemestane reduces the incidence of invasive breast cancer compared with placebo.

Currently: To determine the frequency of serious adverse events for post-menopausal women at high-risk of developing breast cancer who choose to receive 5 years of exemestane as preventative therapy.

Secondary

Previously: (same as is currently listed in PDQ) Currently: To address the Trial Committee and Sponsor's commitment to allow women who are randomized to the MAP.3 trial to receive 5 years of exemestane therapy.

OUTLINE: This study was a randomized, double-blind, placebo-controlled, multicentre study. Protocol-specified analyses were performed in April 2011. The results of these analyses are posted in the Results section. Following the amendment of May 2011, the study is now open-label and all eligible patients are receiving exemestane from participating sites for a total of 5 years. After exemestane is stopped, there is no further follow-up.

PROJECTED ACCRUAL:There were 4560 women from the United States, Canada, Spain and France who took part in this study.

ELIGIBILITY:
* At increased risk of developing breast cancer, due to at least one of the following risk factors:

  * Gail score ≥ 1.66
  * Age ≥ 60 years
  * Prior atypical ductal hyperplasia, lobular hyperplasia, or lobular carcinoma in situ on breast biopsy
  * Prior ductal carcinoma in situ (DCIS) treated with total mastectomy with or without tamoxifen (tamoxifen must have been completed ≥ 3 months prior to randomization)
* No prior DCIS treated with lumpectomy with or without radiation
* No prior invasive breast cancer
* Not BRCA1 or BRCA2 carriers

PATIENT CHARACTERISTICS:

Previous:

* 35 and over
* Female
* Postmenopausal, defined as one of the following:

  * over 50 years of age with no spontaneous menses for at least 12 months before study entry
  * 50 years of age or under with no menses (spontaneous or secondary to hysterectomy) for at least 12 months before study entry AND with follicle-stimulating hormone level within postmenopausal range
  * Underwent prior bilateral oophorectomy
* No other malignancies within the past 5 years except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid tumors with no evidence of disease for ≥ 5 years
* No uncontrolled hypothyroidism or hyperthyroidism
* No major medical or psychiatric illness (including substance and alcohol abuse within the past 2 years) that would preclude study participation or compliance
* Must be accessible for treatment and follow-up
* Willing to complete quality of life questionnaires in either English or French

Current: MAP.3 participants who were randomized to the exemestane arm, are currently receiving exemestane as part of the MAP.3 study and who have not completed 5 years of exemestane.

OR MAP.3 study participants who were randomized to the placebo arm and who have either completed 5 years of study drug or who are still receiving placebo. Note: this applies only to centres that choose to allow placebo "cross-over".

PRIOR CONCURRENT THERAPY:

Previous:

* More than 3 months since prior and no concurrent hormone replacement therapies
* More than 3 months since systemic estrogenic, androgenic, or progestational agents
* More than 3 months since prior and no concurrent hormonal therapies, including, but not limited to the following:

  * Luteinizing-hormone releasing-hormone analogs (e.g., goserelin or leuprolide)
  * Progestogens (e.g., megestrol)
  * Prolactin inhibitors (e.g., bromocriptine)
  * Antiandrogens (e.g., cyproterone acetate)
  * Selective estrogen-receptor modulators (e.g., tamoxifen, toremifene, or raloxifene)
* No investigational drug within 30 days or 5 half lives prior to randomization
* No concurrent endocrine therapy
* No concurrent estrogens, androgens, or progesterones
* Concurrent low dose (≤ 100 mg/day) prophylactic aspirin allowed
* Concurrent bisphosphonates for prevention or treatment of osteoporosis allowed
* No other concurrent medications that may have an effect on study endpoints

Current: There are no prior concurrent therapy restrictions for the amended MAP.3 study.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4560 (Actual)
Dates: Start 2004-12-03 (Actual); Primary Completion 2011-03-25 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (76):
- United States (41):
  - Jefferson Clinic, P.C., Birmingham, Alabama
  - UAB Comprehensive Cancer Center-LNB 301, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of California, San Diego, La Jolla, California
  - University of California at Davis, Sacramento, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Whittingham Cancer Center at Norwalk Hospital, Norwalk, Connecticut
  - The George Washington University, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Georgia Cancer Specialists, Tucker, Georgia
  - John H. Stroger, Jr Hospital of Cook County, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Centre, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Mid-Illinois Hematology and Oncology Associates, Ltd., Normal, Illinois
  - Carle Cancer Centre, Urbana, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Suburban Hospital Cancer Program, Bethesda, Maryland
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hutzel Women's Health Specialists, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Kinston Medical Specialists, Kinston, North Carolina
  - University of Cincinnati, Barrett Cancer Centre, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Abramson Cancer Center of the, Philadelphia, Pennsylvania
  - The Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Fletcher Allen Health Care, Burlington, Vermont
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Univ. of Wisconsin Center for Women's Health and, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (20):
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Meadowlands Family Health Centre, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUM - Pavillon Saint-Luc, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
- France (13):
  - CRLCC - Paul Papin, Angers
  - CHU-Hopital A. Morvan, Brest
  - Centre Francois Baclesse, Caen
  - CHU de Limoges - Hopital Mere Enfant, Limoges
  - CHU - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Rene Gauducheau, Nantes
  - Clinique Hartmann, Neuilly-sur-Seine
  - AP-HP Hopital Tenon, Paris
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave-Roussy, Villejuif
- Puerto Rico (2):
  - Orocovis Medical Center, Orocovis
  - Altamira Family Research Center, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson H, Johnston D, Pater J, Goss P. The National Cancer Institute of Canada Clinical Trials Group MAP.3 trial: an international breast cancer prevention trial. Curr Oncol. 2007 Jun;14(3):89-96. doi: 10.3747/co.2007.117. PMID 17593981
- [Result] Goss PE, Richardson H, Chlebowski R, Johnston D, Sarto GE, Maunsell E, Ingle JN, Ales-Martinez JE. National Cancer Institute of Canada Clinical Trials Group MAP.3 Trial: evaluation of exemestane to prevent breast cancer in postmenopausal women. Clin Breast Cancer. 2007 Dec;7(11):895-900. doi: 10.3816/CBC.2007.n.057. No abstract available. PMID 18269782
- [Result] Moy B, Richardson H, Johnston D, et al.: NCIC CTG MAP.3: enrollment and study drug adherence of ethnic minority women in a breast cancer prevention trial. [Abstract] Breast Cancer Res Treat 106 (1): A-3048, S141-2, 2007.
- [Result] Richardson H, Johnston D, Goss PE, et al.: Participant characteristics on an international NCIC CTG breast cancer prevention trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-1531, 2007.
- [Result] Goss PE, Ingle JN, Alés-Martinez J, Cheung A, Chlebowski RT, Wactawski-Wende J, McTiernan A, Robbins J, Johnson K, Martin L, Winquist E, Sarto G, Garber JE, Fabian CJ, Pujol P, Maunsell E, Farmer P, Gelmon KA, Tu D, Richardson H. Exemestane for primary prevention of breast cancer in postmenopausal women: NCIC CTG MAP.3 - A randomized placebo-controlled clinical trial. J Clin Oncol 29[suppl; abstr LBA504], 2011.
- [Result] Goss PE, Ingle JN, Ales-Martinez JE, Cheung AM, Chlebowski RT, Wactawski-Wende J, McTiernan A, Robbins J, Johnson KC, Martin LW, Winquist E, Sarto GE, Garber JE, Fabian CJ, Pujol P, Maunsell E, Farmer P, Gelmon KA, Tu D, Richardson H; NCIC CTG MAP.3 Study Investigators. Exemestane for breast-cancer prevention in postmenopausal women. N Engl J Med. 2011 Jun 23;364(25):2381-91. doi: 10.1056/NEJMoa1103507. Epub 2011 Jun 4. PMID 21639806
- [Derived] Maunsell E, Goss PE, Chlebowski RT, Ingle JN, Ales-Martinez JE, Sarto GE, Fabian CJ, Pujol P, Ruiz A, Cooke AL, Hendrix S, Thayer DW, Rowland KM, Dube P, Spadafora S, Pruthi S, Lickley L, Ellard SL, Cheung AM, Wactawski-Wende J, Gelmon KA, Johnston D, Hiltz A, Brundage M, Pater JL, Tu D, Richardson H. Quality of life in MAP.3 (Mammary Prevention 3): a randomized, placebo-controlled trial evaluating exemestane for prevention of breast cancer. J Clin Oncol. 2014 May 10;32(14):1427-36. doi: 10.1200/JCO.2013.51.2483. Epub 2014 Apr 7. PMID 24711552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 11, 2004, and March 23, 2010, 4560 women were recruited in medical clinics.
Pre-assignment Details: Eligibility of women was first checked before the randomization to the trial.
Groups:
- Randomization Period: Exemestane; Open-label Extension: Exemestane: one 25 mg tablet daily in am
- Randomization Period: Placebo: one tablet daily in am
Period: Randomization Period
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo | Open-label Extension: Exemestane
Started | 2285 | 2275 | 0
Completed | 2285 (All women randomized were included in the analysis based on intent-to-treat principle.) | 2275 (All women randomized were included in the analysis based on intent-to-treat principle.) | 0
Not Completed | 0 | 0 | 0
Period: Open-label Extension
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo | Open-label Extension: Exemestane
Started | 0 | 0 | 2831
Completed | 0 | 0 | 2831
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo | Total
Number analyzed (Participants) | 2285 | 2275 | 4560
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1458 | 1481 | 2939
  >=65 years | 827 | 794 | 1621
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (7.2) | 63.1 (7.0) | 63.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2285 | 2275 | 4560
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1416 | 1408 | 2824
  France | 9 | 10 | 19
  Canada | 643 | 642 | 1285
  Spain | 217 | 215 | 432

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Serious Adverse Events
Description: Percentage of serious adverse events for women who choose to receive 5 years of exemestane as preventative therapy.
Time Frame: 5 years open-label extension period
Population: Postmenopausal women who were randomized to exemestane in original MAP.3 study and chose to continue to receive exemestane for up to 5 years and those randomized to placebo and decided to start 5 years of exemestane.
Measure: Number (95% Confidence Interval); unit: percentage of women
Groups:
- Open-label Extension: Exemestane: one 25 mg tablet daily in am
  exemestane: one 25 mg tablet daily in am
Arm/Group | Open-label Extension: Exemestane
Number analyzed (Participants) | 2831
percentage of women | 0.0 [0.0 to 0.5]

2. Primary Outcome: Invasive Breast Cancer Incidence (Breast Cancer-Free Survival)
Description: Invasive breast cancer incidence was estimated from the breast cancer-free survival (BCFS) which was calculated for all women from the day of the randomization to the earliest date of diagnosis for invasive breast cancer. Women who died from other causes were censored at the time of death. If a woman did not develop an invasive breast cancer, or died, BCFS was censored on the date of the last day the woman was known alive (LKA), which was the latest of the date of assessment. Women who had breast cancer before study entry were also censored at the time of randomization.
Time Frame: Over randomization period of study (median follow-up 35 months)
Population: intention to treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of cases/follow-up person-yr
Groups:
- Randomization Period: Exemestane: 25 mg of exemestane tablet daily
- Randomization Period: Placebo: Placebo tablet daily
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo
Number analyzed (Participants) | 2285 | 2275
percentage of cases/follow-up person-yr | 0.19 [0.08 to 0.30] | 0.55 [0.36 to 0.73]
Statistical Analysis 1: Comparison: Randomization Period: Exemestane vs Randomization Period: Placebo; The null hypothesis was no difference between two groups. The sample size estimate was based on an assumption of annual invasive breast cancer rate of 0.60% in the placebo group and 0.21% in exemestane group, a relative reduction of 65% with exemestane. To detect this with a two-sided 5% level and 90% power, a total of 38 cases of invasive breast cancer were required, projected to occur when 4560 women were randomly assigned in a 3-year period and then followed for an additional 1.2 years; Test type: Superiority or Other; p = 0.002, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.18 to 0.70]

3. Secondary Outcome: Total Incidence of Invasive and Non-invasive (DCIS) Breast Cancer
Description: It was estimated from the Total Breast Cancer-Free Survival (TBCFS), which was calculated for women who developed invasive or non-invasive (DCIS) breast cancer as the time from the date of randomization to the earliest date of diagnosis for invasive or non-invasive (DCIS) breast cancer. Women who died from other causes were censored at the time of death. Women who had breast cancer before entry were censored at the time of randomization. If a woman did not develop an invasive or non-invasive (DCIS) breast cancer, or died, TBCFS will be censored on the date of last known alive.
Time Frame: Over randomization period of study (median follow-up 35 months)
Population: Intent-to-treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of cases/follow-up person-yr
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo
Number analyzed (Participants) | 2285 | 2275
percentage of cases/follow-up person-yr | 0.35 [0.20 to 0.50] | 0.77 [0.54 to 0.99]
Statistical Analysis 1: Comparison: Randomization Period: Exemestane vs Randomization Period: Placebo; Test type: Superiority or Other; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.27 to 0.79]

4. Secondary Outcome: Incidence of Lobular Carcinoma in Situ, Atypical Ductal Hyperplasia and Atypical Lobular Hyperplasia Events
Time Frame: Over randomization period of study (median follow-up 35 months)
Population: Intent-to-treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of cases/follow-up person-yr
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo
Number analyzed (Participants) | 2285 | 2275
percentage of cases/follow-up person-yr | 0.07 [0.00 to 0.15] | 0.20 [0.08 to 0.32]
Statistical Analysis 1: Comparison: Randomization Period: Exemestane vs Randomization Period: Placebo; Test type: Superiority or Other; p = 0.07, Log Rank; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.11 to 1.12]

5. Secondary Outcome: Number of Clinical Breast Biopsies
Time Frame: Over randomization period of study (median follow-up 35 months)
Population: Women who had at least one clinical breast biopsy
Measure: Median (Full Range); unit: number of clinical breast biopsies
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo
Number analyzed (Participants) | 81 | 118
number of clinical breast biopsies | 1 [1 to 3] | 1 [1 to 3]

6. Secondary Outcome: Incidence of All Clinical Fractures
Time Frame: During protocol treatment over randomization period of study (up to 5 years)
Population: Women who have received treatment
Measure: Number; unit: participants
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo
Number analyzed (Participants) | 2240 | 2248
participants | 149 | 143

7. Secondary Outcome: Incidence of Clinically Relevant Cardiac Events
Description: Events including myocardial infarctions and angina requiring percutaneous transluminal coronary angioplasty or coronary artery bypass graft, fatal and nonfatal strokes and all vascular deaths
Time Frame: During protocol treatment in randomization period (up to 5 years)
Population: Women who received treatment during randomization period
Measure: Number; unit: participants
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo
Number analyzed (Participants) | 2240 | 2248
participants | 106 | 111

8. Secondary Outcome: Incidences of Other Malignancies
Description: Other malignancies includes any other malignancy which is not in breast.
Time Frame: Over randomization period of study (median follow-up 35 months)
Population: Women who have received treatment
Measure: Number; unit: participants
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo
Number analyzed (Participants) | 2240 | 2248
participants | 50 | 42

ADVERSE EVENTS:
Time Frame: Participants were followed for a median of 35 months over randomization period of study for randomization period, and 5 years for open-label extension period
Description: During 5 year open-label extension, only SAE was monitored.
Arm/Group | Randomization Period: Exemestane | Randomization Period: Placebo | Open-label Extension: Exemestane
Serious Adverse Events (participants affected / at risk) | 39/2240 | 26/2248 | 0/2831
Other Adverse Events (participants affected / at risk) | 1963/2240 | 1901/2248 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization Period: Exemestane (N=2240) | Randomization Period: Placebo (N=2248) | Open-label Extension: Exemestane (N=2831)
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Supraven.arrhyth. Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 2 | 3 | 0
Valvular heart disease (Cardiac disorders) | 1 | 0 | 0
Cardiac General - Other (Cardiac disorders) | 2 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0
Endocrine - Other (Endocrine disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Incontinence, anal (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Obstruction, GI Stomach (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
GI - Other (Gastrointestinal disorders) | 3 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Pancreatitis (Hepatobiliary disorders) | 0 | 1 | 0
Infec.w.norm.ANC Upper airway NOS (Infections and infestations) | 1 | 0 | 0
Infection (doc.clin.) Lung (Infections and infestations) | 0 | 1 | 0
Infection - Other (Infections and infestations) | 2 | 1 | 0
ALT (Metabolism and nutrition disorders) | 1 | 1 | 0
AST (Metabolism and nutrition disorders) | 1 | 1 | 0
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 | 0 | 0
Creatinine (Metabolism and nutrition disorders) | 1 | 0 | 0
GGT (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
CNS ischemia (Nervous system disorders) | 7 | 4 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 0 | 1 | 0
Ocular - Other (Eye disorders) | 1 | 0 | 0
Pain Abdomen NOS (General disorders) | 1 | 0 | 0
Pain Back (General disorders) | 1 | 0 | 0
Pain Joint (General disorders) | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Syndromes - Other (General disorders) | 0 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization Period: Exemestane (N=2240) | Randomization Period: Placebo (N=2248) | Open-label Extension: Exemestane (N=0)
hypertension (Cardiac disorders) | 341 | 354 | 0
hot flashes (Endocrine disorders) | 900 | 718 | 0
fatigue (Endocrine disorders) | 525 | 465 | 0
sweating (Endocrine disorders) | 486 | 433 | 0
insomnia (Endocrine disorders) | 230 | 189 | 0
Diarrhea (Gastrointestinal disorders) | 118 | 75 | 0
heartburn (Gastrointestinal disorders) | 332 | 289 | 0
Nausea (Gastrointestinal disorders) | 155 | 122 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 247 | 196 | 0
dizziness (Nervous system disorders) | 189 | 209 | 0
mood alteration or depression (Nervous system disorders) | 236 | 235 | 0
Pain Back (General disorders) | 306 | 222 | 0
pain extremity (General disorders) | 153 | 122 | 0
Pain Joint (General disorders) | 665 | 606 | 0
pain muscle (General disorders) | 147 | 192 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 234 | 266 | 0
vaginal dryness (Reproductive system and breast disorders) | 352 | 343 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No